CLINICAL TRIAL: NCT01525953
Title: Predictors of Survival for Complete Clinical Responders to Definite Chemoradiation or Radiation Therapy for Esophageal Cancer
Brief Title: Complete Clinical Responders to Definite Chemoradiation in Esophageal Cancer : a Survival Analysis
Acronym: CRCRT-EC
Status: Completed | Type: Observational
Sponsor: Centre Oscar Lambret (Other)
Responsible Party: Sponsor
Other Study IDs: CRCRT-EC
Record Dates: First submitted 2012-01-30; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Esophageal Cancer
Keywords: esophageal cancer; radiochemotherapy; prognosis
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Drug Therapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy according to standard
Radiation: Radiotherapy — Radiotherapy according to local standard

SUMMARY:
The aim of this study is to identify prognostic factors for outcome in patients being complete clinical responders with chemoradiation or radiation for esophageal cancer

ELIGIBILITY:
Inclusion Criteria:

* localized or locally advanced esophageal cancer
* patient who underwent definite chemoradiation or radiation
* patient with complete clinical response

Exclusion Criteria:

* metastatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient treated for esophageal cancer in the Northern France Cancer Center from january 1998 to december 2003
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2012-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Identification of prognostic factors for overall survival | From date of treatment until death, assessed up to 10 years
  Correlation between survival and baseline,clinical and treatment characteristics

SECONDARY OUTCOMES:
Patterns of treatment failure | From date of treatment until treatment failure, assessed up to 10 years
  Type of recurrence : local, regional, distant.
Disease-free survival | From date of treatment until progression or death, assessed up to 10 years
  Time between the end of treatment and the occurence of progression

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ADENIS, MD, PhD, Principal Investigator — Centre Oscar Lambret
Locations (1):
- Centre Oscar LAMBRET, Lille, France